CLINICAL TRIAL: NCT00085956
Title: Effects of Arzoxifene on Bone Mineral Density and Endometrial Histology in Postmenopausal Women.
Brief Title: Effects of Arzoxifene on Bone Mass and the Uterus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 8537; H4Z-MC-GJAE
Record Dates: First submitted 2004-06-18; First posted 2004-06-22 (Estimated); Last update posted 2007-03-09 (Estimated); Status verified 2007-03

CONDITIONS: Postmenopausal Bone Loss
MeSH Terms: conditions — Osteoporosis, Postmenopausal | interventions — LY 353381

INTERVENTIONS:
Drug: Arzoxifene
Drug: Placebo

SUMMARY:
The purposes of this study are to determine:

* The effects of arzoxifene on bone mineral density (bone mass) at the spine and hip in postmenopausal women.
* The effects of arzoxifene on the uterus (womb) in postmenopausal women.
* The effects of arzoxifene on blood tests that measure changes in bone rebuilding in postmenopausal women with low bone density.
* The effects of arzoxifene on blood lipids (fats) and other blood markers of heart disease risk.
* The safety of arzoxifene and any side effects that might be associated with its use.

ELIGIBILITY:
Inclusion Criteria:

* Female
* 45 to 60 years of age, inclusive
* At least 2 years since last menstrual cycle
* Intact uterus (womb).

Exclusion Criteria:

* Existing fracture of the spine.
* Bone disorders, other than low bone mass
* History of cancer in the last 5 years. Also, any history, at any time, of breast cancer or cancer of the lining of the uterus.
* Abnormal or unexplained vaginal bleeding.

Ages: 45 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300
Dates: Start 2004-04; Study Completion 2007-02

PRIMARY OUTCOMES:
The effects of arzoxifene on bone mineral density (bone mass) at the spine and hip in postmenopausal women
The effects of arzoxifene on the uterus (womb) in post menopausal women
The safety of arzoxifene and any side effects that might be associated with its use

SECONDARY OUTCOMES:
The effects of arzoxifene on blood tests that measure changes in bone rebuilding in postmenopausal women with low bone density
The effects of arzoxifene on blood lipids (fats) and other blood markers of heart disease
The effects of arzoxifene on breast density

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY(1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559), Mon - Fri 9 AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Diego, California, United States

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com